CLINICAL TRIAL: NCT00088400
Title: A Phase III Multicenter Study of Intratumoral/Interstitial Therapy With TransMID Compared to Best Standard of Care in Patients With Progressive and/or Recurrent, Non-Resectable Glioblastoma Multiforme
Brief Title: Comparison of TransMID vs Standard Treatment of Cancerous Brain Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040244; 04-N-0244
Record Dates: First submitted 2004-07-23; First posted 2004-07-26 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Glioblastoma
Keywords: Transferrin; Brain Tumor; Convection; Immunotherapy; Targeted Protein Toxin; Glioblastoma Multiforme; GBM
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Tf-CRM107

INTERVENTIONS:
Drug: TransMID

SUMMARY:
Study Objectives:

Primary Objective:

To evaluate the efficacy of intratumoral/interstitial therapy with TransMID compared to best standard of care in patients with progressive and/or recurrent, non-resectable glioblastoma multiforme.

Secondary Objectives:

To assess the safety of intratumoral/interstitial therapy with TransMID compared to best standard of care in patients with progressive and/or recurrent, non-resectable glioblastoma multiforme.

To evaluate possible differences in efficacy and/or safety with TransMID associated with differing degrees of transferrin receptor expression in tumor tissue and serum anti-diphtheria toxin antibody titer levels.

Study Design:

Multicenter, open label, randomized study comparing TransMID with a chemotherapeutic regimen considered to be best standard of care and consisting of either nitrosureas, platinum compounds, temozolomide, procarbazine or PCV (procarbazine, lomustine (CCNU) & vincristine). A planned interim analysis of the primary efficacy endpoint will be conducted after approximately 50 percent of the required events have been observed.

DETAILED DESCRIPTION:
Study Objectives:

Primary Objective:

To evaluate the efficacy of intratumoral/interstitial therapy with TransMID compared to best standard of care in patients with progressive and/or recurrent, non-resectable glioblastoma multiforme.

Secondary Objectives:

To assess the safety of intratumoral/interstitial therapy with TransMID compared to best standard of care in patients with progressive and/or recurrent, non-resectable glioblastoma multiforme.

To evaluate possible differences in efficacy and/or safety with TransMID associated with differing degrees of transferrin receptor expression in tumor tissue and serum anti-diphtheria toxin antibody titer levels.

Study Design:

Multicenter, open label, randomized study comparing TransMID with a chemotherapeutic regimen considered to be best standard of care and consisting of either nitrosureas, platinum compounds, temozolomide, procarbazine or PCV (procarbazine, lomustine (CCNU) & vincristine). A planned interim analysis of the primary efficacy endpoint will be conducted after approximately 50 percent of the required events have been observed.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients will be included in the study if they meet all of the following criteria:

1. Male or female at least 18 years of age.
2. Histological results confirming GBM are available.
3. Progressive GBM (greater than or equal to 25 percent increase in contrast enhanced tumor CSA compared to the nadir or smallest previous measured CSA) and/or recurrent GBM after conventional treatment, including surgery (biopsy or debulking surgery) and/or radiation therapy and/or chemotherapy.
4. Pre-study MRIs used to determine current progression and/or recurrence of GBM are available to the Investigator and for independent confirmation of progression and/or recurrence.
5. Patient is not considered a candidate for resection.
6. If female of child-bearing potential, a reliable method of contraception must be combined with a negative pregnancy test before entering the study (female patients must be willing to use contraception for 2 months after the last treatment with TransMID (Trademark)). Male patients must be willing to use a barrier method of contraception for up to 2 months after the last treatment with TransMID (Trademark)
7. Able and willing to follow instructions and comply with the protocol.
8. Provide written informed consent prior to participation in the study.
9. Karnofsky Performance Scale Score 70-100.
10. Tumor characteristics:

    i) must be unifocal; and

ii) must be unilateral and supratentorial; and

iii) lesion must have a diameter (on contrast-enhanced MRI) greater than or equal to 1.0 cm and less than or equal to 4.0 cm.

EXCLUSION CRITERIA:

Patients will be excluded from the study if they meet any of the following criteria:

1. Anticipated life expectancy of less than 3 months.
2. Infratentorial or intraventricular tumors.
3. Presence of satellite tumors.
4. Chemotherapy within 30 days prior to study entry or nitrosureas or Mitomycin-C containing therapy within 42 days prior to study entry.
5. Radiotherapy or stereotactic (gamma knife) radiosurgery within 90 days prior to study entry.
6. Tumor surgery, tumor debulking or other neurosurgery within 30 days prior to study entry.
7. Previous administration of TransMID (Trademark)
8. Previous enrollment in this study.
9. Regional therapy including administration of biodegradable polymer wafers containing carmustine within 90 days prior to study entry or brachytherapy within 12 calendar months prior to study entry.
10. Significant liver function impairment-(total bilirubin greater than 2.0 mg/dl or 34.2 mircomol/L; AST or ALT greater than 3 times the upper limit of normal).
11. Significant renal impairment (serum creatinine greater than 1.7 mg/dL or 150 micromol/L).
12. Coagulopathy (prothrombin time [PT] or activated partial thromboplastin time [APTT] greater than 1.5 times control).
13. Thrombocytopenia (platelet count less than 100 x 10(3)/micro-L or 100 x 10(9)/L).
14. Granulocytopenia (absolute neutrophil count (ANC), less than 1 x 10(3)/micro-L or 1.0 x 10(9)/L).
15. Severe acute infection.
16. Medical condition that is considered an unacceptable anesthetic risk.
17. Evidence of a mass effect on CT or MRI with more than a 5 mm midline shift and/or nausea, vomiting, reduced level of consciousness or clinically significant papilledema.
18. Nursing or pregnant females. A pregnancy test will be performed on all females who are of child-bearing potential.
19. Use of any investigational product and/or participation in another clinical research study within the last 30 days prior to study entry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-07; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ameri A, Poisson M, Chen QM, Delattre JY. Treatment of recurrent malignant supratentorial gliomas with the association of procarbazine, thiotepa and vincristine: a phase II study. J Neurooncol. 1993 Jul;17(1):43-6. doi: 10.1007/BF01054273. PMID 8120571
- [Background] Angelova-Gateva P. Iron transferrin receptors in rat and human cerebrum. Agressologie. 1980;21(1):27-30. No abstract available. PMID 6263123
- [Background] Bobo RH, Laske DW, Akbasak A, Morrison PF, Dedrick RL, Oldfield EH. Convection-enhanced delivery of macromolecules in the brain. Proc Natl Acad Sci U S A. 1994 Mar 15;91(6):2076-80. doi: 10.1073/pnas.91.6.2076. PMID 8134351